CLINICAL TRIAL: NCT01610076
Title: Pilot Study to Determine Effectiveness and Acceptance of a Code Status Video in the ICU
Brief Title: Code Status Video in the Intensive Care Unit: Video Assisted Patient Education
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kianoush B. Kashani, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-003628
Record Dates: First submitted 2012-01-31; First posted 2012-06-01 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Critical Illness
Keywords: Code Status; Do not resuscitate (DNR); Do not intubate (DNI); CPR; Cardiopulmonary resuscitation; video; advanced directives
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Video - Control (No Intervention): This group does not watch the 10 minute "code status" video before having the knowledge base video administered.
- Code Status Video (Experimental): This group views a 10 minute video about "code status" prior to knowledge base survey administration
  Interventions: Other: Code Status Video

INTERVENTIONS:
Other: Code Status Video — 10 minute video about "Code Status"
  Arms: Code Status Video

SUMMARY:
This is a single-center, randomized control trial of a code status video as an educational tool in the intensive care unit. Subjects are stratified by patient or surrogate and are randomized to either watch an educational video on code status or not watch the video. They are then asked knowledge base questions regarding code status as well as questions pertaining to comfort regarding code status. Participants randomized to watch the video are also asked questions related to acceptance of the video.

DETAILED DESCRIPTION:
After randomization subjects will be divided into control group and intervention group that will receive video tutorial. All subjects will have unlimited access to printed brochures about Advance Directives available at our institution. Use of those materials will be left to their discretion of patients, surrogates and health care professionals involved in patients care. This study was conducted in the medical ICU of tertiary medical center.

Educational video tutorial to cardiovascular resuscitation, defibrillation, endotracheal intubation and mechanical ventilation. Video presents illustrations of resuscitation performed on actors. It informs about the risk, benefits and statistical outcomes of Cardiopulmonary resuscitation (CPR).

Immediately after admission to ICU patients or their health care surrogates were asked to participate in the study. The time between admission and enrollment varied depending on patient's needs and feasibility of conducting research. Upon enrollment subjects were stratified into two groups. One was composed of patients participating in education and testing and another composed of health care surrogates participating on patient's behalf. Those groups were further divided to intervention group that received video education and control group. Stratified randomization occurred according to computer generated list which will be followed for duration of the study. Patients in all four groups had access to printed brochures about Advance Directives. Those pamphlets were available at the admission desk and at the nursing stations. All participants were tested from their knowledge of the code status and related terminology. Subjects randomized to the control group were tested immediately after obtaining consent. Subject from intervention group were tested immediately after video education. Test was administered by the investigator in the format of interview. Completion of the questionnaire took <10 minutes. Questionnaire contained 17 testing questions. Questionnaire was validated and piloted prior to actual trial.

Satisfaction from education as well as level of discomfort caused by participation in the study were assessed with numeric scales. Following the interview all participants were asked if they would like to discuss Code Status preferences with physician taking care of them. If so, response were noted and appropriate services will be notified immediately. If patients were unable to consent to the study or participate in video education and testing, their health care surrogates were allowed to participate on behalf of the patient. Person giving the consent participated as a subject. Participation of health care proxy were tracked in the collected data. Patient's medical record number was used as personalized code for all the subjects including health care surrogates.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18 and older admitted to the medical intensive care unit

Exclusion Criteria:

* Institutionalized status (prisoners)
* Pregnancy
* A priori decided comfort care measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2010-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kianoush B Kashani, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Hofmann JC, Wenger NS, Davis RB, Teno J, Connors AF Jr, Desbiens N, Lynn J, Phillips RS. Patient preferences for communication with physicians about end-of-life decisions. SUPPORT Investigators. Study to Understand Prognoses and Preference for Outcomes and Risks of Treatment. Ann Intern Med. 1997 Jul 1;127(1):1-12. doi: 10.7326/0003-4819-127-1-199707010-00001. PMID 9214246
- [Background] Wenger NS, Phillips RS, Teno JM, Oye RK, Dawson NV, Liu H, Califf R, Layde P, Hakim R, Lynn J. Physician understanding of patient resuscitation preferences: insights and clinical implications. J Am Geriatr Soc. 2000 May;48(S1):S44-51. doi: 10.1111/j.1532-5415.2000.tb03140.x. PMID 10809456
- [Background] Teno JM, Hakim RB, Knaus WA, Wenger NS, Phillips RS, Wu AW, Layde P, Connors AF Jr, Dawson NV, Lynn J. Preferences for cardiopulmonary resuscitation: physician-patient agreement and hospital resource use. The SUPPORT Investigators. J Gen Intern Med. 1995 Apr;10(4):179-86. doi: 10.1007/BF02600252. PMID 7790978
- [Background] von Gunten CF, Ferris FD, Emanuel LL. The patient-physician relationship. Ensuring competency in end-of-life care: communication and relational skills. JAMA. 2000 Dec 20;284(23):3051-7. doi: 10.1001/jama.284.23.3051. PMID 11122596

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Video - Control | Code Status Video
Started | 103 | 105
Completed | 100 | 100
Not Completed | 3 | 5
Not completed — Technical issue with video | 0 | 1
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Video - Control | Code Status Video | Total
Number analyzed (Participants) | 103 | 105 | 208
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [47 to 73] | 58 [44 to 73] | 60 [45 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 53 | 105
  Male | 51 | 52 | 103
Region of Enrollment [Number; unit: participants]
  United States | 103 | 105 | 208

OUTCOME MEASURES:

1. Primary Outcome: 12 Question Resuscitation Status Survey (Question 4 Has 4 Sub-questions)
Description: 12 question (question 4 has 4 sub-questions) survey previously validated to determine knowledge level about resuscitation status with total score on the scale of 0-15. Possible scores ranged from 0 to 15, with higher scores representing increased medical knowledge.
  The CPR knowledge survey assesses a participants basic understanding of cardiopulmonary resuscitation (CPR). The survey consisted of 12 questions with one point being awarded for each correct response. Question four had a total of four possible correct answers. Thus the scores on the scale of 0-15 points is designed, with higher scores representing increased knowledge.
Time Frame: after admission to ICU, approx one hour
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | No Video - Control | Code Status Video
Number analyzed (Participants) | 103 | 105
points | 6.5 [5 to 9.75] | 9 [6 to 12]

2. Secondary Outcome: Participant Reported Comfort With Video Intervention
Description: Patient's were surveyed about "How comfortable were you watching the video?"
Time Frame: immediately after intervention
Population: Patient's surveyed about
Measure: Number; unit: participants
Arm/Group | Code Status Video
Number analyzed (Participants) | 100
participants
  Very Comfortable Watching the Video | 75
  Somewhat Comfortable Watching the video | 24
  Not Comfortable watching the video | 1

3. Secondary Outcome: Perception of Utility of Video
Description: Participants were surveyed, "How helpful was this video in helping you understand your options?" There possible answers were provided:
  Very helpful Somewhat helpful Not helpful
Time Frame: immediately after intervention
Measure: Number; unit: participants
Arm/Group | Code Status Video
Number analyzed (Participants) | 100
participants
  Very helpful | 70
  Somewhat helpful | 28
  Not helpful | 2

4. Secondary Outcome: Willingness to Recommend Video to Other Patients
Description: Participants were surveyed, "Would you recommend this video to other patients?" Three options were provided:
  Definitely recommend Probably recommend Do not recommend
Time Frame: immediately after intervention
Measure: Number; unit: participants
Arm/Group | Code Status Video
Number analyzed (Participants) | 100
participants
  Definitely recommend | 70
  Probably recommend | 29
  Do not recommend | 1

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the course of the accrual. As investigators believed that watching a video could not cause significant physical damage following the post-video interview, the follow up ended for each individual patient.
Arm/Group | No Video - Control | Code Status Video
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/105
Other Adverse Events (participants affected / at risk) | 0/103 | 0/105

LIMITATIONS AND CAVEATS:
In this study the patient outcomes were not addressed as the primary outcome was patient and family knowledge of CPR.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No